CLINICAL TRIAL: NCT00390377
Title: A Study to Evaluate a Test for the Diagnosis of Breast Cancer Using X-Ray Diffraction of Hair Fibres.
Brief Title: Use of Hair to Diagnose Breast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fermiscan Ltd (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: FT240-2006
Record Dates: First submitted 2006-10-17; First posted 2006-10-19 (Estimated); Last update posted 2006-10-19 (Estimated); Status verified 2006-10

CONDITIONS: Breast Cancer
Keywords: x-ray diffraction; hair; breast cancer; synchrotron
MeSH Terms: conditions — Breast Neoplasms

INTERVENTIONS:
Procedure: Cutting scalp hair

SUMMARY:
This study aims to perform x-ray diffraction analysis of blinded hair samples from women with a documented health status, to validate the previous findings of James et al who described that x-ray diffraction patterns of human hair can distinguish samples from healthy subjects from those of diseased subjects, specifically those suffering from breast cancer.

The primary hypothesis is that x-ray diffraction of hair can be used to distinguish hair from patients with confirmed breast cancer from subjects without detectable breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Adult women (aged >20) who are undergoing mammography, and
* Who are willing and able to provide informed consent; and
* Who have usable scalp hair

Exclusion Criteria:

* Women with a history of breast cancer ever or other cancers (excluding non-melanoma skin cancer and CIN: cervical intra-epithelial neoplasia) within 5 years.

Min Age: 20 Years | Sex: Female
Age Groups: Adult, Older Adult
Enrollment: 240
Dates: Start 2006-10

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Shnier, MBBS, FRACR, Principal Investigator — Symbion Health; Gary Corino, BSc, Study Director — Fermiscan Ltd
Locations (1):
- St George Private Hospital, Sydney, New South Wales, Australia

REFERENCES:
- [Background] James V, Corino G, Robertson T, Dutton N, Halas D, Boyd A, Bentel J, Papadimitriou J. Early diagnosis of breast cancer by hair diffraction. Int J Cancer. 2005 May 10;114(6):969-72. doi: 10.1002/ijc.20824. PMID 15645416
- [Background] James V, Kearsley J, Irving T, Amemiya Y, Cookson D. Using hair to screen for breast cancer. Nature. 1999 Mar 4;398(6722):33-4. doi: 10.1038/17949. No abstract available. PMID 10078527
- [Background] Meyer P, James VJ. Experimental confirmation of a distinctive diffraction pattern in hair from women with breast cancer. J Natl Cancer Inst. 2001 Jun 6;93(11):873-5. doi: 10.1093/jnci/93.11.873. No abstract available. PMID 11390537
- [Background] James VJ. The traps and pitfalls inherent in the correlation of changes in the fibre diffraction pattern of hair with breast cancer. Phys Med Biol. 2003 Jan 21;48(2):L5-9; discussion L11-3. doi: 10.1088/0031-9155/48/2/101. PMID 12587913
- [Background] Kimura M, Tanaka N, Kimura Y, Miyake K, Kitaura T, Fukuchi H. Pharmacokinetic interaction of zonisamide in rats. Effect of other antiepileptics on zonisamide. J Pharmacobiodyn. 1992 Nov;15(11):631-9. doi: 10.1248/bpb1978.15.631. PMID 1289498
- [Background] James V. False-positive results in studies of changes in fiber diffraction of hair from patients with breast cancer may not be false. J Natl Cancer Inst. 2003 Jan 15;95(2):170-1. doi: 10.1093/jnci/95.2.170. No abstract available. PMID 12529353